CLINICAL TRIAL: NCT01798628
Title: A Phase 1, Single Dose, Open-Label, Three-Period, Crossover Study to Determine the Effect of Food on the Pharmacokinetics of Abiraterone Acetate in Healthy Male Subjects
Brief Title: A Study to Determine the Effect of Food on the Pharmacokinetics of Abiraterone Acetate in Healthy Male Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016960; COU-AA-009 (Other: Cougar Biotechnology, Inc.)
Record Dates: First submitted 2012-10-22; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Abiraterone acetate; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence ABC (Experimental)
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate
- Sequence ACB (Experimental)
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate
- Sequence BAC (Experimental)
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate
- Sequence BCA (Experimental)
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate
- Sequence CAB (Experimental)
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate
- Sequence CBA (Experimental)
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate

INTERVENTIONS:
Drug: Treatment A: abiraterone acetate — 1000 mg (4 x 250 mg tablets) taken by mouth as a single dose administered after a high-fat meal
Drug: Treatment B: abiraterone acetate — 1000 mg (4 x 250 mg tablets) taken by mouth as a single dose after a low-fat meal
Drug: Treatment C: abiraterone acetate — 1000 mg (4 x 250 mg tablets) taken by mouth as a single dose administered in the fasted state

SUMMARY:
The purpose of this study is to determine the effect of food on the pharmacokinetics (how the drug concentrations change over time) of abiraterone acetate 1000 mg when administered as a single dose in healthy male volunteers.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known), randomized (treatment sequences will be assigned by chance) study of a single dose of abiraterone acetate 1000 mg administered orally (by mouth) in approximately 36 healthy male participants under fasted and fed conditions. Three doses of abiraterone acetate will be administered with a 7-day washout period between each dose. The total study duration for each participant will be 21 days. Participants will be randomized to one of six treatment sequences (ABC, ACB, BAC, BCA, CAB, CBA): Treatment A = abiraterone acetate 1000 mg administered after a high-fat meal; Treatment B = abiraterone acetate 1000 mg administered after a low-fat meal; Treatment C = abiraterone acetate 1000 mg administered in the fasted state. No food will be ingested for 4 hours post-dose. Participants will be confined at the clinical research unit from the day prior to dosing until clinic discharge on the day following dosing in each treatment period. Serial pharmacokinetic samples will be collected and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* In good general health as determined by no clinically significant findings on medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory measurements
* Body mass index within 18 kg/m2 to 32 kg/m2, inclusive
* Non-tobacco users
* Clinical laboratory values within protocol-defined parameters
* Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]),and negative human immunodeficiency virus (HIV) antibody screens
* Negative test for selected drugs of abuse
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Significant history or manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological or psychiatric disorder, as determined by the Principal Investigator
* History or presence of an abnormal electrocardiogram
* History of stomach or intestinal surgery resection that would potentially alter absorption and/or excretion of orally administered drugs
* Screening serum total testosterone of <200 ng/dL
* History of hypersensitivity reaction to the study drug, related compounds or excipients used in the formulation
* Receipt of an investigational drug within 5 half-lives or 30 days prior to Day -1, whichever is longer
* Abnormal diet during the 30 days prior to Day 1
* Donation of blood or significant loss of blood within 56 days or plasma within 14 days prior to Day -1
* Planned donation of blood or plasma from Screening through Study Completion, Day 21
* Receipt of blood products within 2 months prior to Day 1
* History of protocol-defined alcohol abuse
* Known or suspected use of illicit drugs within the last year
* Use of any medication on a chronic basis
* Use of any prescription medications/products or over-the-counter non-prescription preparations within 5 half-lives or 7 days prior to Day -1 unless deemed acceptable by the Sponsor
* Consumption of alcohol-containing foods or beverages within 24 hours prior to the first Check-in (Day -1)
* Unwillingness to abstain from alcohol consumption from Day -1 to Study Completion (Day21)
* Consumption of caffeine-containing or grapefruit-containing foods or beverages within 72 hours prior to Day -1
* Unwillingness to abstain from caffeine-containing or grapefruit-containing foods or beverages from Day -1 through Study Completion (Day21)
* Presence of sexual dysfunction or any medical condition that would affect sexual function
* Unwillingness to refrain from strenuous exercise from 48 hours prior to Day -1 and for the duration of the study
* Presence of any condition that, in the opinion of the Investigator, would limit the participant's ability to complete and/or participate in this study
* Unwillingness to refrain from using any tobacco or nicotine-containing products during screening and throughout the study to Study Completion (Day 21)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of abiraterone | Within 1 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Time to maximum concentration of abiraterone | Within 1 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Area under the concentration-time curve from time 0 to the last measurable concentration of abiraterone | Within 1 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Area under the concentration-time curve extrapolated to infinity of abiraterone | Within 1 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Apparent plasma terminal elimination rate constant of abiraterone | Within 1 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Apparent terminal elimination half-life of abiraterone | Within 1 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose

SECONDARY OUTCOMES:
Number of participants affected by an adverse event | Up to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.